CLINICAL TRIAL: NCT04422873
Title: The Impact of Coronavirus (COVID-19) Restrictions on Wellbeing, Quality of Life and Physical Activity in People With End-stage Renal Disease, Currently Dialysing In-centre Versus at Home in the UK and Their Experience of Telemedicine
Brief Title: The Impact of COVID-19 on Dialysis Users
Status: Completed | Type: Observational
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); University of Reading (Other)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Other Study IDs: 004
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: End Stage Renal Disease; Sars-CoV2
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- in-centre: Currently dialysing in-centre
- home: Currently dialysing at home

SUMMARY:
To understand the impact of COVID-19 restrictions on the wellbeing, quality of life and physical activity of people with end-stage renal disease, currently dialysing in-centre versus at home in the UK and their experience of telemedicine.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is an infectious disease caused by a newly discovered coronavirus. Most people infected with the COVID-19 virus will experience mild-to-moderate respiratory illness, however, some older people and those with underlying medical problems are more likely to develop serious illness.

One group who are particularly vulnerable at this time is people with chronic kidney disease (CKD). Of this group, particularly at risk are those at the more severe end of the disease spectrum [end stage renal disease (ESRD], who rely on renal replacement therapy (RRT), in the form of dialysis, to do the job of the kidneys. The investigators currently have a programme of clinical research investigating the impact of home versus in-hospital RRT, using both qualitative (IRAS: 264200) and quantitative approaches (IRAS: 254251). A key focus of this work is to explore determinants of wellbeing, function and overall quality of life that are linked to dialysis modality.

On Monday 23rd March, the UK Government imposed significant restrictions with regards to human movement, for at least three weeks (recently extended to at least 6 weeks) to try and reduce the risk of the COVID-19 disease spreading within the UK. These included: only shopping for basic necessities; one form of exercise a day, such as a walk, run or cycle; travel for specific medical needs; those travelling to and from work, where this is absolutely necessary and it cannot be done from home.

This is an interesting time, since it is usually observed that people who dialysis at home (i.e. home haemodialysis) typically have more freedom to go out, as they do not have the thrice weekly commute to a renal clinic, which is a burden itself, to then undergo ~4 hours of dialysis at the unit. People who dialyse at home are now isolating entirely and in charge of their own treatment, resulting in very little contact with others. The Wessex Kidney Centre has, however, implemented remote clinics and has been trialling an application to assess patient-reported outcome measures (PROMs) as part of its ongoing programme of research. Those dialysing in-centre however, continue to have contact with medical staff in person thrice weekly and are forced to break isolation and go into a clinical setting.

Through the proposed study, the research team will capture patients' experience during this unique and unprecedented time, in order to guide practice moving forwards and identify potential areas for intervention. More specifically, the purpose of this study is to understand the impact of COVID-19 restrictions on the wellbeing, quality of life and physical activity of people with end-stage renal disease, currently dialysing in-centre versus at home in the UK and their experience of telemedicine. This information may be used to help us better support individuals in the future and investigate the feasibility of telemedicine in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Willing and able to undertake the interview process
* Able to give informed consent

Exclusion Criteria:

* Age < 18 years
* Does not provide written informed consent
* Any neurological/psychiatric diagnoses
* Lack of fluency in English
* Individuals who have commenced RRT within three months of the study start date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with advanced ESRD (eGFR < 15 mL/min/1.73m2) will be recruited into this study.
  Persons falling into two distinct categories will be approached:
  1. ESRD on ICHD
  2. ESRD on HHD
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of the effect of COVID-19 restrictions on patients' well-being, quality of life and physical activity and sedentary behaviours | Day 1
  Participants will be asked during a qualitative interview about the effect of COVID-19 restrictions on their; well-being, quality of life and physical activity and sedentary behaviours

SECONDARY OUTCOMES:
Thematic analysis of qualitative interview exploring patients' experiences of telemedicine during the COVID-19 restrictions in the UK | Day 1
  Participants will be asked during a qualitative interview about their perceptions and experiences of telemedicine

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Health and Exercise Science, Portsmouth, Outside the United States Or Canada, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Transcripts will not be uploaded to repositories